CLINICAL TRIAL: NCT05323656
Title: A Phase 2, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Setanaxib, When Administered With Pembrolizumab, in Patients With Recurrent or Metastatic SCCHN
Brief Title: A Study of Setanaxib Co-Administered With Pembrolizumab in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck (SCCHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calliditas Therapeutics Suisse SA (Industry)
Responsible Party: Sponsor
Organization: Calliditas Therapeutics AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSN000400
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Squamous Cell Carcinoma of Head and Neck; Setanaxib; Pembrolizumab; SCCHN; Keytruda
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — setanaxib; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Setanaxib 1600 mg and Pembrolizumab 200 mg (Experimental): Participants will be administered setanaxib at a dose of 1600 mg/day for the up to 24-month double-blind treatment period.
  Participants will also be administered Pembrolizumab 200 mg intravenously every 3 weeks.
  Interventions: Drug: Setanaxib; Biological: Pembrolizumab
- Placebo and Pembrolizumab 200 mg (Active Comparator): Participants will be administered placebo for the up to 24-month double-blind treatment period.
  Participants will also be administered Pembrolizumab 200 mg intravenously every 3 weeks.
  Interventions: Biological: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Setanaxib — Oral tablets, 400 mg per tablet
  Arms: Setanaxib 1600 mg and Pembrolizumab 200 mg
Biological: Pembrolizumab — 200 mg IV infusion
  Other Names: Keytruda
Drug: Placebo — Oral tablets
  Arms: Placebo and Pembrolizumab 200 mg

SUMMARY:
The primary objective of this study is to compare the change in tumour size per Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1) in recurrent or metastatic SCCHN patients treated with setanaxib and pembrolizumab versus patients treated with placebo and pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years, inclusive, at the time of informed consent.
* Willing and able to give informed consent and to comply with the requirements of the study.
* Histologically- or cytologically-confirmed diagnosis of SCCHN that is recurrent or metastatic with or without nodal involvement, and with or without metastatic spread, and is not eligible for surgical resection.
* Candidates for first-line treatment for pembrolizumab for recurrent or metastatic SCCHN, at the discretion of the investigator.
* A positive CAFs level (defined as CAFs level in tumours ≥5%), performed at a central laboratory, with fresh tumour biopsy taken during or within 30 days prior to the Screening Period. If available, suitable archival tissue (taken within 6 months prior to the Screening Visit and where the patient has received no further anti-cancer therapy during this 6-month period) can be used to assess tumour CAFs level and determine patient eligibility.
* Measurable disease, in accordance with RECIST v1.1, and with tumour accessible and of sufficient volume for pre-treatment and on-treatment biopsy.
* Combined positive score (CPS) ≥1, as determined on the archival or fresh tumour biopsy taken during or within 30 days prior to the Screening Period.
* HPV status known at randomisation.
* Life expectancy of at least 6 months in the judgment of the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ and bone marrow function within 35 days of starting study treatment. Criteria "a" to "c" cannot be met in patients with ongoing or recent (within 14 days of screening test) transfusions or who require ongoing growth factor support:

  1. Absolute neutrophil count ≥1,000/mm3 (≥ 1.0×109/L).
  2. Platelet count ≥100,000/mm3 (≥ 100×109/L).
  3. Haemoglobin ≥9 g/dL, in the absence of transfusions for at least 2 weeks. Patients requiring ongoing transfusions or growth factor support to maintain haemoglobin ≥ 9g/dL are not eligible.
  4. Total bilirubin ≤1.5×upper limit of normal (ULN) (if associated with liver metastases or Gilbert's disease, ≤3×ULN).
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN.
  6. Serum creatinine ≤2.0 mg/dL or creatinine clearance ≥40 mL/min (measured or calculated according to the method of Cockcroft and Gault).
* Female patients of childbearing potential must use a highly effective method of contraception to prevent pregnancy for ≥4 weeks before randomisation and must agree to continue strict contraception up to 120 days after the last dose of IMP or pembrolizumab, whichever is the later.

  1. For the purposes of this study, women of childbearing potential are defined as "fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy."
  2. Postmenopausal state is defined as no menses for 12 months without an alternative medical cause. In female patients who are not using hormonal contraception or hormonal replacement therapy but with suspected menopause and less than 12 months of amenorrhea, a high follicle stimulating hormone (FSH) level in the postmenopausal range will be required at Screening to confirm a postmenopausal state. Confirmation with more than one FSH measurement is required.
  3. Highly effective contraception is defined as methods that can achieve a failure rate of less than 1% per year when used consistently and correctly.
* Female patients of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline/Randomisation before dosing.
* Male patients with female partners of childbearing potential must be willing to use a condom and require their partner to use an a highly effective contraceptive method.
* Male patients must refrain from donating sperm, and female patients must refrain from donating eggs, from Baseline until 120 days after the last dose of IMP or pembrolizumab, whichever is the later.

Exclusion Criteria:

* Diagnosis of immunosuppression or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at doses not to exceed 10 mg/day of prednisone or equivalent. Steroids as premedication for hypersensitivity reactions due to radiographic contrast agents are allowed.
* Anti-cancer mAb treatment within 4 weeks prior to study Day 1.
* Chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 (radiation therapy can be allowed for palliative therapy of bone metastasis only).
* Not recovered from AEs Grade 2 or greater (except for alopecia) due to previously administered agents.
* Treatment with any investigational agent within 12 weeks of Screening Visit or 5 half-lives of the IMP (if known), whichever is longer, or current enrolment in an interventional clinical study.
* Prior treatment with setanaxib or participation in a previous setanaxib clinical study.
* Prior treatment with pembrolizumab.
* Known additional malignancy that is progressing or requires active treatment excepting basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer that has undergone potentially curative therapy, or malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IMP and of low potential risk for recurrence.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Active autoimmune disease requiring systemic treatment within the past 3 months or documented history of clinically severe autoimmune disease, or syndrome that requires systemic steroids or immunosuppressive agents. The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia.
  2. Any chronic skin condition that does not require systemic therapy.
  3. Patients with coeliac disease controlled by diet alone.
* Any evidence of current interstitial lung disease or pneumonitis, or a prior history of interstitial lung disease or non-infectious pneumonitis requiring high-dose glucocorticoids.
* Active infection requiring systemic therapy.
* Known human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B or C infection. Patients with a past or resolved hepatitis B virus infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of hepatitis B surface antigen [HBsAg]) are eligible provided the hepatitis virus DNA test is negative. Patients positive for hepatitis C antibody are eligible only if polymerase chain reaction (PCR) is negative for hepatitis C virus RNA. Patients with ongoing anti-viral therapy with potent inhibitors of cytochrome P450 (CYP) 3A4 are not eligible. Testing for HIV is only required if clinically indicated and is not mandatory for this study.
* Serious chronic gastrointestinal conditions associated with diarrhoea.
* History of significant haematological problems, such as blood dyscrasias requiring treatment, aplastic anaemia, myelodysplastic syndrome, or leukaemia.
* Surgery (eg, stomach bypass) or medical condition that might significantly affect absorption of medicines (as judged by the investigator).
* A positive pregnancy test or breastfeeding for female patients.
* Evidence of any of the following cardiac conduction abnormalities: a QTc Fredericia interval >450 milliseconds for male patients or >470 milliseconds for female patients. Patients with a second- or third-degree atrioventricular block are to be excluded.
* TSH >ULN at Screening.
* Unstable cardiovascular disease as defined by any of the following:

  1. Unstable angina within 6 months prior to Screening
  2. Myocardial infarction, coronary artery bypass graft surgery, or coronary angioplasty within 6 months prior to Screening
  3. Cerebrovascular accident within 6 months prior to Screening
  4. New York Heart Association Class III or IV heart failure
* Presence of any laboratory abnormality or condition that, in the opinion of the investigator, could interfere with or compromise a patient's treatment, assessment, or compliance with the protocol and/or study procedures.
* Any other condition that, in the opinion of the investigator, constitutes a risk or contraindication for the participation of the patient in the study, or that could interfere with the study objectives, conduct, or evaluation.
* Use of medications known to be potent CYP3A4 inhibitors or inducers, or potent uridine diphosphate (UDP)-glucuronosyltransferase 1A9 (UGT1A9) inhibitors or inducers, within 21 days prior to IMP administration.
* Legal incapacity or limited legal capacity.
* Psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Patients who are unable to provide informed consent, are incarcerated or unable to follow protocol requirements.
* Previous randomisation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2025-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (5):
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Washington University School of Medicine Center for Advanced Medicine, St Louis, Missouri
- France (8):
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Grand Est
  - Centre de Lutte contre le Cancer - Centre Oscar Lambret, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire Amiens-Picardie - Site Sud, Amiens, Picardie
  - Ramsay Health Clinic Belharra, Bayonne
  - Hôpital Saint-André, Bordeaux
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
- Medizinische Hochschule Hannover, Hanover, Lower Saxony, Germany
- Italy (2):
  - Azienda Socio-Sanitaria Territoriale Santi Paolo e Carlo - Ospedale San Paolo Polo Universitario, Milan, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Poland (2):
  - Centrum Onkologii Im. Prof. F. Łukaszczyka w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie-Państwowy Instytut Badawczy O. w Gliwicach, Gliwice, Silesian Voivodeship
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (2):
  - The Royal Marsden Hospital - London, London, England
  - The Royal Marsden Hospital Head and Neck Unit, Sutton, England

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Setanaxib 1600 mg and Pembrolizumab 200 mg: Participants will be administered setanaxib at a dose of 1600 mg/day for the up to 24-month double-blind treatment period.
  Participants will also be administered Pembrolizumab 200 mg intravenously every 3 weeks.
  Setanaxib: Oral tablets, 400 mg per tablet
  Pembrolizumab: 200 mg IV infusion
- Placebo and Pembrolizumab 200 mg: Participants will be administered placebo for the up to 24-month double-blind treatment period.
  Participants will also be administered Pembrolizumab 200 mg intravenously every 3 weeks.
  Placebo: Oral tablets
  Pembrolizumab: 200 mg IV infusion
Period: Overall Study
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Started | 27 | 28
Completed | 1 | 1
Not Completed | 26 | 27
Not completed — Still On-Treatment | 6 | 6
Not completed — Progressive Disease | 15 | 14
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Clinical disease progression | 0 | 1
Not completed — Patient and Investigator decision | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10) | 65.0 (10.54) | 64.8 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 22 | 18 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 17 | 14 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 22 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 6 | 16
Human papillomavirus (HPV) Status [Count of Participants; unit: Participants]
  Positive | 5 | 5 | 10
  Negative | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Best Percentage Change in Tumour Size
Description: Defined as the best percentage change from Baseline in the sum of diameters of target lesions, as assessed by RECIST v1.1.
Time Frame: Baseline to at least 15 weeks and up to 51 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 26 | 28
Percentage change from baseline | -7.88 (9.323) | -12.93 (8.977)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Null hypothesis: the mean best percentage change in the tumour size between the treatment groups are the same. With 25 patients per treatment group, using a 2-sided t-test, there will be 85% power to detect a 20% mean difference between the treatment groups in best percentage change in tumour size, with an estimated standard deviation of 30% and a 2 sided alpha of 20%; Test type: Superiority; p = 0.7008, ANCOVA; LS Mean Difference = 5.05, 80% CI 2-sided [-11.98 to 22.0], Standard Error of Mean 13.077 — The LS Mean difference is for the Setanaxib Group minus the Placebo Group

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as time from randomisation to the first documented disease progression per RECIST v1.1 or death due to any cause, whichever occurs first.
Time Frame: Baseline up to approximately 21 months
Population: Full Analysis Set
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 27 | 28
days | 151 [125 to 229] | 87 [65 to 117]
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Null hypothesis: The risk for progression, as defined by RECIST v1.1, is the same between treatment groups. If the true hazard ratio is 0.5, approximately 38 progression events as defined by RECIST v1.1 will be required to have > 80% power to demonstrate a statistically significant difference in PFS with 2-sided p<0.2; Test type: Superiority; p = .1023, Regression, Cox; Hazard Ratio (HR) = 0.58, 80% CI 2-sided [0.38 to 0.89]

3. Secondary Outcome: Change From Baseline in Cancer-associated Fibroblasts (CAFs) Level in Tumour Tissue
Description: Changes within treatment groups (ie, across paired tissue samples) and between treatment groups summarized both descriptively and as adjusted mean difference between treatment groups.
Time Frame: Baseline up to approximately 9 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: % positivity of tumour stromal component
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 10
% positivity of tumour stromal component
  Baseline | 58.13 (37.006) | 52.00 (23.357)
  Week 9 | 50.50 (31.023) | 36.50 (30.373)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Null Hypothesis: Mean difference in postbaseline CAF levels does not differ between treatment groups. ANCOVA model is on postbaseline CAFs level with a fixed factor for treatment and a covariate for baseline; Test type: Superiority; p = 0.2986, ANCOVA — a priori threshold for significance (0.2) not met; LS Mean Difference = 9.5, 80% CI 2-sided [-2.3 to 21.3], Standard Error of Mean 8.89 — The LS Mean difference is for the Setanaxib Group minus the Placebo Group

4. Secondary Outcome: Change From Baseline in the Number of Cluster of Differentiation 8 (CD8+) Tumour Infiltrating Lymphocytes (TILs) in Tumour Tissue
Description: as for outcome 3
Time Frame: Baseline up to approximately 9 weeks
Population: Full Analysis Set)
Measure: Mean (Standard Deviation); unit: cells/High Power Field (HPF)
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 11 | 8
cells/High Power Field (HPF)
  Baseline | 18.13 (8.901) | 21.34 (19.789)
  Week 9 | 41.14 (34.535) | 38.30 (26.553)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Null Hypothesis: Mean difference in postbaseline CD8+ TILs does not differ between treatment groups. ANCOVA model is on postbaseline CD8+ TILs level with a fixed factor for treatment and a covariate for baseline; Test type: Superiority; p = 0.5918, ANCOVA; LS Mean Difference = 6.83, 80% CI 2-sided [-9.86 to 23.52], Standard Error of Mean 12.48 — The LS Mean difference is for the Setanaxib Group minus the Placebo Group

5. Secondary Outcome: Change From Baseline in the Number of Regulatory T-cells in Tumour Tissue
Description: as for outcome 3
Time Frame: Baseline up to approximately 9 weeks
Measure: Mean (Standard Deviation); unit: cells/High Power Field (HPF)
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 11 | 8
cells/High Power Field (HPF)
  Baseline | 9.75 (9.955) | 24.36 (27.104)
  Week 9 | 21.14 (22.879) | 30.16 (38.866)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Null Hypothesis: Mean difference in postbaseline number of regulatory T-cells in tumour tissue does not differ between treatment groups. ANCOVA model is on postbaseline number of regulatory T-cells in tumour tissue level with a fixed factor for treatment and a covariate for baseline; Test type: Superiority; p = 0.2135, ANCOVA; LS Mean Difference = 10.84, 80% CI 2-sided [-0.34 to 22.02], Standard Error of Mean 8.37 — The LS Mean difference is for the Setanaxib Group minus the Placebo Group

6. Secondary Outcome: Overall Response Rate (ORR)
Description: Proportion of the patients who have a complete response (CR) or partial response (PR) per RECIST v1.1 will be used to access ORR.
Time Frame: Baseline up to approximately 12 months
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 27 | 28
Participants
  Complete Response | 1 | 0
  Partial Response | 8 | 9
  Stable Disease | 10 | 5
  Progressive Disease | 7 | 14
  Not Evaluable | 1 | 0

7. Secondary Outcome: Duration of Response (DoR)
Description: The minimum time when CR or PR is first observed to the time of progression of disease (PD) or death will be used to access DoR.
Time Frame: Baseline up to approximately 12 months
Population: Full Analysis Set
Measure: Number (80% Confidence Interval); unit: days
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 27 | 28
days
  Duration of Response 25% Percentile | 170 [64 to NA] — Insufficient number of participants with events | 46 [43 to 79]
  Duration of Response 50% Percentile | NA [170 to NA] — Insufficient number of participants with events | 79 [49 to NA] — Insufficient number of participants with events
  Duration of Response 75% Percentile | NA [170 to NA] — Insufficient number of participants with events | 300 [79 to NA] — Insufficient number of participants with events

8. Secondary Outcome: Disease Control Rate (DCR)
Description: Proportion of the patients in whom the best overall response is determined as CR, PR, or stable disease (SD) per RECIST v1.1 will be used to access DCR.
Time Frame: Baseline up to approximately 12 months
Population: Full Analysis Set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 27 | 28
percentage of participants | 70.4 [54.5 to 82.5] | 50 [35.2 to 64.8]

9. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from randomisation to death due to any cause. Patients without documented death at the time of the final analysis will be censored at the date of the last follow-up.
Time Frame: Baseline up to 12 months
Population: Full Analysis Set
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 27 | 28
percentage of participants
  3 Months | 96 [91.3 to 100] | 79 [68.6 to 88.5]
  6 Months | 92 [85.6 to 99.0] | 68 [56.5 to 79.2]
  9 Months | 88 [79.1 to 96.3] | 58 [45.9 to 71.0]
  12 Months | 46 [19.4 to 72.5] | 42 [26.0 to 58.2]
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; No formal test of significance undertaken; Test type: Superiority; Hazard Ratio (HR) = 0.448, 80% CI 2-sided [0.24 to 0.85]

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Any clinically significant abnormalities in vital signs, physical examination, clinical laboratory tests (including biochemistry, hematology, urinalysis, and thyroid function), or 12- lead electrocardiogram (ECG) results will be recorded as Adverse Events (AEs).
Time Frame: Baseline up to approximately 21 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 27 | 28
Participants | 27 | 26

11. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: AESI include Anaemia and Hypothyroidism.
Time Frame: Baseline up to approximately 21 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 27 | 28
Participants | 5 | 5

12. Secondary Outcome: Levels of Programmed Death-ligand 1 (PD-L1) Expression in Tumour Tissue
Description: Combined Positive Score (CPS) is a scoring method that predicts response to pembrolizumab in patients with cancer defined as the number of PD-L1-staining cells (tumor cells, lymphocytes, and macrophages) relative to the total number of viable tumor cells. A higher CPS score indicates an increased likelihood to respond to pembrolizumab treatment. It was hypothesized based on the mode of action of setanaxib that there would be an increased immunological response and therefore an increase in PD-L1 in tumor tissue.
  Changes within treatment groups (ie, across paired tissue samples) and between treatment groups summarized both descriptively and as adjusted mean difference between treatment groups.
Time Frame: Baseline up to approximately 9 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 11 | 7
ratio
  Baseline | 19.73 (29.408) | 13.14 (25.149)
  Week 9 | 42.27 (37.641) | 18.57 (15.999)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Null Hypothesis: Mean difference in postbaseline PD-L1 combined positive score (CPS) does not differ between treatment groups. ANCOVA model is on postbaseline PD-L1 CPS with a fixed factor for treatment and a covariate for baseline. Threshold for statistical significance = 0.2; Test type: Superiority; p = 0.0782, ANCOVA; The LS Mean difference is for the Setanaxib Group minus the Placebo Group; Mean Difference (Final Values) = 17.76, 80% CI 2-sided [5.17 to 30.36], Standard Error of Mean 9.4

13. Secondary Outcome: Change From Baseline in CAFs Cell Type Abundance Based on Gene Expression Profiles
Description: Digital cytometry was carried out using CIBERSORTx. This estimates cell type abundance based on gene expression profiles in bulk RNA-Seq data. The abundance of myofibroblastic CAF were enumerated using a custom signature matrix based on gene expression profiles derived from annotated SCCHN scRNA-Seq data.
  CIBERSORTx Absolute Abundance ratio is calculated by the median expression level of all genes in the signature matrix divided by the median expression level of all genes in the mixture (bulk RNA-Seq data for the sample). This produces a score that quantitatively measures the overall abundance of each cell type using gene expression profiles.
Time Frame: Baseline up to approximately 9 weeks
Population: Full Analysis Set with paired observations
Measure: Mean (Standard Deviation); unit: CIBERSORTx Absolute Abundance ratio
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 11
CIBERSORTx Absolute Abundance ratio
  Screening | 0.87 (0.880) | 0.74 (0.787)
  Week 9 | 0.98 (0.990) | 0.56 (0.581)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Within group test of hypothesis that screening and week 9 values are equal; Test type: Other; p = 0.22, Wilcoxon signed rank test; Mean Difference (Net) = 0.11, Standard Deviation 0.578
Statistical Analysis 2: Comparison: Placebo and Pembrolizumab 200 mg; Within group test of hypothesis that screening and week 9 values are equal; Test type: Other; p = 0.20, Wilcoxon signed rank test; Mean Difference (Net) = -.18, Standard Deviation 0.395

14. Secondary Outcome: Change From Baseline in CD8+ TILs Cell Type Abundance Based on Gene Expression Profiles
Description: Digital cytometry was carried out using CIBERSORTx. This estimates cell type abundance based on gene expression profiles in bulk RNA-Seq data. The abundance of tumor-infiltrating lymphocytes (TILs) were enumerated using a custom signature matrix based on gene expression profiles derived from annotated SCCHN scRNA-Seq data.
  CIBERSORTx Absolute Abundance ratio is calculated by the median expression level of all genes in the signature matrix divided by the median expression level of all genes in the mixture (bulk RNA-Seq data for the sample). This produces a score that quantitatively measures the overall abundance of each cell type using gene expression profiles.
Time Frame: Baseline up to approximately 9 weeks
Population: Full Analysis Set with paired observations
Measure: Mean (Standard Deviation); unit: CIBERSORTx Absolute Abundance ratio
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 11
CIBERSORTx Absolute Abundance ratio
  Screening | 0.03 (0.030) | 0.04 (0.044)
  Week 9 | 0.07 (0.063) | 0.02 (0.033)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg; Within group test of hypothesis that screening and week 9 values are equal; Test type: Other; p = 0.037, Wilcoxon signed rank test; Mean Difference (Net) = 0.05, Standard Deviation 0.069
Statistical Analysis 2: Comparison: Placebo and Pembrolizumab 200 mg; Within group test of hypothesis that screening and week 9 values are equal; Test type: Other; p = 0.123, Wilcoxon signed rank test; Mean Difference (Net) = -0.02, Standard Deviation 0.039

15. Secondary Outcome: Change From Baseline in Regulatory T-cell Abundance Based on Gene Expression Profiles
Description: Digital cytometry was carried out using CIBERSORTx. This estimates cell type abundance based on gene expression profiles in bulk RNA-Seq data. The abundance of regulatory T-cells were enumerated using a custom signature matrix based on gene expression profiles derived from annotated SCCHN scRNA-Seq data.
  CIBERSORTx Absolute Abundance ratio is calculated by the median expression level of all genes in the signature matrix divided by the median expression level of all genes in the mixture (bulk RNA-Seq data for the sample). This produces a score that quantitatively measures the overall abundance of each cell type using gene expression profiles.
Time Frame: Baseline up to approximately 9 weeks
Population: Full Analysis Set with paired observations
Measure: Mean (Standard Deviation); unit: CIBERSORTx Absolute Abundance ratio
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 11
CIBERSORTx Absolute Abundance ratio
  Screening | 0.01 (0.012) | 0.02 (0.033)
  Week 9 | 0.01 (0.016) | 0.03 (0.054)
Statistical Analysis 1: Comparison: Setanaxib 1600 mg and Pembrolizumab 200 mg vs Placebo and Pembrolizumab 200 mg; Within group test of hypothesis that screening and week 9 values are equal; Test type: Other; p = 0.41, Wilcoxon signed rank test; Mean Difference (Net) = 0.01, Standard Deviation 0.017
Statistical Analysis 2: Comparison: Placebo and Pembrolizumab 200 mg; Within group test of hypothesis that screening and week 9 values are equal; Test type: Other; p = 0.11, Wilcoxon signed rank test; Mean Difference (Net) = 0.01, Standard Deviation 0.023

16. Secondary Outcome: Area Under The Concentration-time Curve Over a 24-hour Period at Steady State (AUC[0-24]-ss) of Setanaxib
Time Frame: Baseline, Week 3, week 9, week 24, week 51
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h*mL-¹
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg
Number analyzed (Participants) | 27
ug*h*mL-¹ | 240.41 (28.86)

17. Secondary Outcome: Area Under The Concentration-time Curve Over a 24-hour Period at Steady State (AUC24-ss) of GKT138184
Time Frame: Baseline, Week 3, week 9, week 24, week 51
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h*mL-¹
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg
Number analyzed (Participants) | 27
ug*h*mL-¹ | 50.2 (41.49)

18. Secondary Outcome: Minimum Plasma Concentration at Steady State (Cmax-ss) of Setanaxib
Time Frame: Baseline, Week 3, week 9, week 24, week 51
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*mL-¹
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg
Number analyzed (Participants) | 27
ug*mL-¹ | 2.14 (85.71)

19. Secondary Outcome: Minimum Plasma Concentration at Steady State (Cmin-ss) of GKT138184
Time Frame: Baseline, Week 3, week 9, week 24, week 51
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*mL-¹
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg
Number analyzed (Participants) | 27
ug*mL-¹ | 0.76 (68.98)

20. Secondary Outcome: Maximum Plasma Concentration at Steady State (Cmax-ss) of Setanaxib
Time Frame: Baseline, Week 3, week 9, week 24, week 51
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*mL-¹
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg
Number analyzed (Participants) | 27
ug*mL-¹ | 26.24 (24.84)

21. Secondary Outcome: Maximum Plasma Concentration at Steady State (Cmax-ss) of GKT138184
Time Frame: Baseline up to approximately 26 months
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*mL-¹
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg
Number analyzed (Participants) | 27
ug*mL-¹ | 3.74 (34.33)

ADVERSE EVENTS:
Time Frame: Reporting of AEs began when the patient had provided informed consent and continued up to 28 days after the last IMP administration, up to 27 months.
Description: Patients were monitored for death also after the adverse event collection period, until approximately 38 progression events as defined by RECIST v1.1 had occurred in the study.
Arm/Group | Setanaxib 1600 mg and Pembrolizumab 200 mg | Placebo and Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 6/27 | 13/28
Serious Adverse Events (participants affected / at risk) | 8/27 | 10/28
Other Adverse Events (participants affected / at risk) | 27/27 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setanaxib 1600 mg and Pembrolizumab 200 mg (N=27) | Placebo and Pembrolizumab 200 mg (N=28)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 (3)
Herpes simplex (Infections and infestations) | 1 (1) | 0
Pneumonia (Infections and infestations) | 1 (1) | 0
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 0
Lipase increased (Investigations) | 1 (1) | 0
Troponin I increased (Investigations) | 1 (1) | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0
Asthenia (Gastrointestinal disorders) | 0 | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Hypotension (Vascular disorders) | 1 (1) | 0
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Setanaxib 1600 mg and Pembrolizumab 200 mg (N=27) | Placebo and Pembrolizumab 200 mg (N=28)
Asthenia (General disorders) | 11 (15) | 9 (14)
Fatigue (General disorders) | 5 (6) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Implant site extravasation (General disorders) | 2 (4) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2)
Xerosis (General disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (10) | 5 (13)
Nausea (Gastrointestinal disorders) | 7 (9) | 5 (6)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (8)
Vomiting (Gastrointestinal disorders) | 4 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (6)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Skin Lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 6 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (6) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 4 (13) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (9) | 2 (7)
Weight decreased (Investigations) | 3 (3) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 9 (11) | 5 (6)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT05323656/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT05323656/SAP_001.pdf